CLINICAL TRIAL: NCT04683211
Title: Evaluation of Iodine Supplementation in Women With Pregnancy Associated With Gestational Diabetes
Acronym: IODIAB
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: IDRCB 2020-A02570-39
Record Dates: First submitted 2020-12-17; First posted 2020-12-24 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Gestational Diabetes
Keywords: Iodine intake; iodine supplementation; gestational diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Evaluation of iodine supplementation — survey of iodine supplementation

SUMMARY:
Iodine supplementation during pregnancy is recommended by the high health authority and by the World Health Organization during pregnancy. We would like to know if this supplementation is prescribed in a manner consistent with the recommendations in women diagnosed with gestational diabetes.

DETAILED DESCRIPTION:
Physiological iodine requirements are increased in pregnant women, from 150 μg / day to 250 μg / day. The iodine intake is assessed by the iodine concentration in the urine, the target of which in pregnant women is ioduria between 150 and 250 μg / l. The general French population is not deficient in iodine according to the national nutrition health study in 2006-2007, with a median ioduria of 136 μg / l (therefore greater than 100 μg / l) for all elderly adults aged 18-74. However, according to French studies, the median ioduria of pregnant women is between 50 and 100 μg / l, which suggests a moderate iodine deficiency. To maintain euthyroidism, the mother must increase her T4 production by 40- 50% (10-150%), which requires an additional iodine intake of 150-250 μg / d The thyroid contains a reserve of iodine, but this is depleted during pregnancy in the absence of supplementation. Our study therefore aims to assess the amount of iodine supplementation prescribed in pregnant women diagnosed with gestational diabetes because this group of patients benefit from early specialized care for their pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* pregnant woman with gestational diabetes
* age ≥ 18 years
* subject informed of the study and not having opposed it.

Exclusion Criteria:

* already known pathology of the thyroid

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with gestational diabetes
Study Population: Women with gestational diabetes
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
Iodine supplementation | Day 0
  µg/day

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France

IPD SHARING:
Plan to Share IPD: No